CLINICAL TRIAL: NCT04798586
Title: A PHASE I, OPEN LABEL STUDY TO EVALUATE THE SAFETY AND PHARMACOKINETIC OF PF 06863135, A B CELL MATURATION ANTIGEN (BCMA) CD3 BISPECIFIC ANTIBODY, AS A SINGLE AGENT IN JAPANESE PARTICIPANTS WITH RELAPSED/REFRACTORY ADVANCED MULTIPLE MYELOMA
Brief Title: MAGNETISMM-2: Study of Elranatamab (PF-06863135) in Japanese Participants With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1071002
Record Dates: First submitted 2021-03-01; First posted 2021-03-15 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-05

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Elranatamab (PF-06863135) (Experimental): BCMA-CD3 bispecific antibody
  Interventions: Drug: Elranatamab (PF-06863135)

INTERVENTIONS:
Drug: Elranatamab (PF-06863135) — BCMA-CD3 bispecific antibody

SUMMARY:
The purpose of this study is to confirm the safety and tolerability of elranatamab (PF-06863135) in Japanese participants with relapsed or refractory MM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (IMWG criteria)
* Measurable disease, as defined by at least 1 of the following

  1. Serum myeloma (M) protein ≥0.5 g/dL (5 g/L)
  2. Urine M protein ≥200 mg/24 h
  3. Serum free light chain (FLC) >100 mg/L (10 mg/dL) with abnormal kappa:lambda ratio
* Participants must have progressed on or been intolerant of at least 3 prior therapies including proteasome inhibitor, IMID drug and anti-CD38 antibody, either in combination or as a single agent
* ECOG PS 0, 1 or 2. PS 3 is permitted if PS is due solely to bone pain
* Adequate bone marrow, hematological, kidney and liver function
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade 1
* Not pregnant and willing to use contraception

Exclusion Criteria:

* POEMS syndrome
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ
* History of active autoimmune disorders
* Any form of primary immunodeficiency
* History of severe immune-mediated adverse event with prior immunomodulatory treatment
* Stem cell transplant within 12 weeks prior to enrollment
* Active graft versus host disease other than Grade 1 skin involvement, or that requiring immunosuppressive treatment
* Requirement for systemic immune suppressive medication
* Active, uncontrolled bacterial, fungal, or viral infection, including HBV, HCV, known HIV or AIDS related illness and SARS-CoV2
* Previous administration with an investigational drug within 4 weeks or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer)
* Known or suspected hypersensitivity to component of elranatamab (PF-06863135), murine and bovine products
* Live attenuated vaccine within 4 weeks

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Japan (2):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Lon HK, Hibma J, Jiang S, Sullivan S, Vandendries E, Skoura A, Wang D, Elmeliegy M. Population Exposure-Response Efficacy Analysis of Elranatamab (PF-06863135) in Patients with Multiple Myeloma. Target Oncol. 2025 Sep;20(5):803-819. doi: 10.1007/s11523-025-01168-y. Epub 2025 Aug 18. PMID 40826257
- [Derived] Elmeliegy M, Viqueira A, Vandendries E, Hickman A, Conte U, Irby D, Hibma J, Lon HK, Piscitelli J, Soltantabar P, Skoura A, Jiang S, Wang D. Dose Optimization of Elranatamab to Mitigate the Risk of Cytokine Release Syndrome in Patients with Multiple Myeloma. Target Oncol. 2025 Mar;20(2):349-359. doi: 10.1007/s11523-025-01134-8. Epub 2025 Feb 25. PMID 40000533
- [Derived] Iida S, Ito S, Yokoyama H, Ishida T, Nagai Y, Handa H, Ito S, Kamei Y, Nakamura M, Suzuki K. Elranatamab in Japanese patients with relapsed/refractory multiple myeloma: results from MagnetisMM-2 and MagnetisMM-3. Jpn J Clin Oncol. 2024 Sep 4;54(9):991-1000. doi: 10.1093/jjco/hyae068. PMID 38794892
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4 participants were screened and assigned to study treatment.
Groups:
- Elranatamab: Participants received an initial priming dose of 600 microgram per kilogram elranatamab subcutaneously on Cycle 0 Day 1 (7 days prior to Cycle 1 Day 1). During treatment cycle, participants were administered 1000 microgram per kilogram elranatamab weekly during each cycle (each cycle was of 3 weeks).
Period: Overall Study
Arm/Group | Elranatamab
Started | 4
Completed | 2
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all enrolled participants who received at least 1 dose of study intervention.
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data cannot be reported due to low enrollment in one category and would lead to risk of re-identification of participants.
  Male | NA — Data cannot be reported due to low enrollment in one category and would lead to risk of re-identification of participants.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following: Treatment Emergent Adverse Events (AEs) occurring in Cycle 0 and Cycle 1 (total 4 weeks): Grade (G) 4 neutropenia lasting greater than (>)7 days; febrile neutropenia (absolute neutrophil count [ANC] less than (<)1,000 per millimeter cube (/mm^3) with single temperature >38.3 degree Celsius (deg C), or sustained temperature of greater than or equal to (>=) 38deg C for >1 hour [h]); G>=3 neutropenia with infection; G4 thrombocytopenia (unless the baseline count was >=25,000/mm^3 and <50,000/mm^3, in which case G4 thrombocytopenia was to be accompanied by >=G2 bleeding), Platelet count <10,000/mm^3 was considered a DLT irrespective of other factors; G3 thrombocytopenia with >=G2 bleeding; G4 AEs; G3 AE >=5 days despite optimal supportive care (except AEs attributed to cytokine release syndrome [CRS]); G3 CRS (except CRS that have not been maximally treated or improved to <=G1 within 48h); confirmed drug induced liver injury.
Time Frame: Up to 4 weeks
Population: Per Protocol Analysis Set included all enrolled participants who had at least 1 dose of study intervention and either experienced DLT or did not have major treatment deviations during the DLT observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (SAEs), Treatment Emergent Treatment Related AEs and Treatment Emergent Treatment Related SAEs
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs included both serious and all non-serious adverse events. An SAE was defined as any untoward medical occurrence that, at any dose resulted in any of the following outcomes: death; life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; or that was considered as an important medical event. A TEAE was defined as an AE that first occurred from the first dose of the study intervention until 90 days after the last dose or the day before starting a new anticancer therapy, whichever occurred first. Treatment related AEs and SAEs were defined as AEs and SAEs which was related to the treatment.
Time Frame: From first dose of study intervention and up to 90 days after last dose or start of new anticancer therapy (maximum of 65.1 weeks of treatment)
Population: SAS included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Participants
  TEAEs | 4
  Treatment Emergent SAEs | 3
  Treatment Emergent Treatment Related AEs | 4
  Treatment Emergent Treatment Related SAEs | 3

3. Secondary Outcome: Number of Participants With Grade 3 or 4, Grade 5 TEAEs and Treatment Related TEAEs Based on Common Terminology Criteria for Adverse Events (CTCAE) Version 5 Except for CRS and ICANS Graded According to ASTCT Grading Criteria 2019
Description: CTCAEv5.0 G3:severe/clinically significant;G4:life-threatening;G5:death.ASTCT CRS G3:temp>=38degC,hypotension required vasopressor with/without vasopressin and/or hypoxia required high-flow nasal cannula,facemask,nonrebreather mask or venturi mask;G4:temp>=38degC,hypotension required multiple vasopressors(excluding vasopressin)and/or hypoxia required positive pressure;G5:death.ICANS G3:ICE score0-2,awakens only to tactile stimulus,clinical seizure focal/generalized resolves rapidly or nonconvulsive seizures on electroencephalography resolve with intervention,focal/local edema on neuroimaging;G4:ICEscore 0(unarousable unable to perform ICE),unarousable or requires vigorous/repetitive tactile stimuli to arouse,stupor/coma,life-threatening prolonged seizure(>5 min),repetitive clinical/electrical seizure without return to baseline,deep focal motor weakness,diffuse cerebral edema on neuroimaging,decerebrate/decorticate posturing,cranial nerve VI palsy,papilledema,Cushing's triad;G5:death.
Time Frame: as for outcome 2
Population: SAS included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Participants
  Grade 3 or 4 TEAEs | 2
  Grade 5 TEAEs | 2
  CRS events | 4
  ICANS events | 0

4. Secondary Outcome: Number of Participants With Shift From Grade Less Than or Equal to (<=) 2 at Baseline to Grade 3 or 4 Post -Baseline in Hematology Parameters by NCI CTCAE v 5.0
Description: Hematology parameters that were assessed included: Anemia, Lymphocyte count decreased, Neutrophil count decreased, Platelet count decreased, White blood cell decreased. Abnormalities were graded based on National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 - Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening.
Time Frame: as for outcome 2
Population: SAS included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Participants
  Anemia | 2
  Lymphocyte count decreased | 4
  Neutrophil count decreased | 3
  Platelet count decreased | 0
  White blood cell decreased | 3

5. Secondary Outcome: Number of Participants With Shift From Grade Less Than or Equal to (<=) 2 at Baseline to Grade 3 or 4 Post -Baseline in Chemistry Parameters by NCI CTCAE v 5.0
Description: Chemistry parameters that were assessed included: Alanine aminotransferase increased, Alkaline phosphatase increased, Aspartate aminotransferase increased, Blood bilirubin increased, Creatinine increased, Hypercalcemia, Hyperkalemia, Hypermagnesemia, Hypernatremia, Hypoalbuminemia, Hypocalcemia, Hypoglycemia, Hypokalemia, Hypomagnesemia, Hyponatremia. Abnormalities were graded based on CTCAE version 5.0- Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening.
Time Frame: as for outcome 2
Population: SAS included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Participants
  Alanine aminotransferase increased | 0
  Alkaline phosphatase increased | 0
  Aspartate aminotransferase increased | 0
  Blood bilirubin increased | 0
  Creatinine increased | 0
  Hypercalcemia | 0
  Hyperkalemia | 0
  Hypermagnesemia | 0
  Hypernatremia | 0
  Hypoalbuminemia | 0
  Hypocalcemia | 0
  Hypoglycemia | 0
  Hypokalemia | 1
  Hypomagnesemia | 0
  Hyponatremia | 0

6. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Elranatamab
Time Frame: Cycle 0: from Cycle 0 Day 1 (pre dose to the next dose of study intervention) [maximum of 9 days]; Cycle 1: from Cycle 1 Day 1 (pre dose to the next dose of study intervention) [maximum of 9 days]
Population: Pharmacokinetic parameter analysis population was defined as all enrolled participants treated who did not have protocol deviations influencing PK assessment and had sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Micrograms per milliliter
  Cycle 0 Day1 | 4.382 (33)
  Cycle 1 Day 1 | 8.846 (39)

7. Secondary Outcome: Time to Maximum Concentration (Tmax) of Elranatamab
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: Days
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Days
  Cycle 0 Day 1 | 7.00 [2.96 to 8.00]
  Cycle 1 Day 1 | 2.98 [2.08 to 5.98]

8. Secondary Outcome: Area Under the Concentration-time Profile From Time Zero to the Time Tau (AUCtau) of Elranatamab
Description: Area under the concentration-time profile from time zero to the time tau where the dosing interval (tau = 1 week). AUCtau was determined using the linear/log trapezoidal method.
Time Frame: as for outcome 6
Population: Pharmacokinetic parameter analysis population was defined as all enrolled participants treated who did not have protocol deviations influencing PK assessment, and had sufficient information to estimate at least 1 of the PK parameters of interest. Here, 'Number Analyzed' signifies participants evaluable at specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*day per milliliter
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Microgram*day per milliliter
  Cycle 0 Day 1 | 21.16 (42)
  Cycle 1 Day 1: number analyzed (Participants) | 2
  Cycle 1 Day 1 | NA (NA) — It was planned that data would not be summarized when there were less than 3 evaluable measurements. Data of individual participants cannot be reported due to risk of re-identification of participants.

9. Secondary Outcome: Pre-dose Trough Serum Concentrations After Multiple Doses of Elranatamab
Time Frame: At pre-dose on Day 1 of Cycle 0, 3, 4, 5, 6, 7, 8, 12, 16; at pre-dose on Days 1, 8, 15 of Cycle 1 and 2
Population: Pharmacokinetic concentration population was defined as all enrolled participants who were treated and had at least 1 analyte concentration. Here, 'Number Analyzed' signifies participants evaluable at specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Microgram per milliliter
  Cycle 0 Day1: Predose | NA (NA) — Summary statistics are not presented if Number of observations Above Lower limit of Quantification (NALQ) = 0 or more than 50% of the concentration data were missing at a particular time point.
  Cycle 1 Day1: Predose | 4.267 (18)
  Cycle 1 Day8: Predose | 8.326 (28)
  Cycle 1 Day15: Predose | 12.32 (34)
  Cycle 2 Day1: Predose | 13.40 (27)
  Cycle 2 Day8: Predose | 16.26 (43)
  Cycle 2 Day15: Predose | 17.83 (45)
  Cycle 3 Day1: Predose | 19.75 (49)
  Cycle 4 Day1: Predose | 21.68 (35)
  Cycle 5 Day1: Predose | 21.71 (43)
  Cycle 6 Day1: Predose | 23.99 (34)
  Cycle 7 Day1: Predose | 18.03 (87)
  Cycle 8 Day1: Predose | 24.27 (51)
  Cycle 12 Day1: Predose: number analyzed (Participants) | 3
  Cycle 12 Day1: Predose | 21.30 (41)
  Cycle 16 Day1: Predose: number analyzed (Participants) | 1
  Cycle 16 Day1: Predose | NA (NA) — Summary statistics are not presented if NALQ = 0 or more than 50% of the concentration data were missing at a particular time point.

10. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) of Elranatamab
Description: 'A participant was considered ADA positive if baseline titer was missing or negative and participant had >=1 post-treatment positive titer, or positive titer at baseline and had a >=4-fold increase in titer from baseline in >=1 post-treatment sample.
Time Frame: From the date of first dose up to maximum of 65.1 weeks of treatment
Population: Immunogenicity analysis set included all enrolled participants who received at least one dose of study treatment and had at least one sample tested for ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Participants | 2

11. Secondary Outcome: Titers of ADA
Description: Titers of ADA at specified timepoints were reported in this outcome measure.
Time Frame: Cycle1 Day1, Cycle1 Day15, Cycle2 Day1, Cycle3 Day1, Cycle4 Day1, Cycle6 Day1, Cycle8 Day1, Cycle12 Day1, Cycle16 Day1, End of treatment (maximum of 65.1 weeks of treatment)
Population: Immunogenicity analysis set included all enrolled participants who received at least one dose of study treatment and had at least one sample tested for ADA. Here, 'Number of Participants Analyzed' signifies ADA positive participants with at least one evaluable sample. 'Number Analyzed' signifies participants with non-missing ADA titers at each time point.
Measure: Mean (Standard Deviation); unit: Titers
Arm/Group | Elranatamab
Number analyzed (Participants) | 2
Titers
  Cycle1 Day1: number analyzed (Participants) | 0
  Cycle1 Day15: number analyzed (Participants) | 0
  Cycle2 Day1: number analyzed (Participants) | 0
  Cycle3 Day1: number analyzed (Participants) | 0
  Cycle4 Day1: number analyzed (Participants) | 0
  Cycle6 Day1: number analyzed (Participants) | 0
  Cycle8 Day1: number analyzed (Participants) | 0
  Cycle12 Day1: number analyzed (Participants) | 1
  Cycle12 Day1 | NA (NA) — Data cannot be reported due to risk of re-identification of participant.
  Cycle16 Day1: number analyzed (Participants) | 0
  End of treatment: number analyzed (Participants) | 1
  End of treatment | NA (NA) — Data cannot be reported due to risk of re-identification of participant.

12. Secondary Outcome: Number of Participants With Neutralizing Antibodies (NAb)
Description: A participant was considered NAb positive if baseline titer was missing or negative and participant had >=1 post-treatment positive titer, or positive titer at baseline and had a >=4-fold increase in titer from baseline in >=1 post-treatment sample.
Time Frame: From the date of first dose up to maximum of 65.1 weeks of treatment
Population: Immunogenicity analysis set included all enrolled participants who received at least one dose of study treatment and had at least one sample tested for ADA. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Elranatamab
Number analyzed (Participants) | 2
Participants | 0

13. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With Objective Response
Description: ORR:% of participants with best overall response; confirmed stringent complete response(sCR),CR, very good partial response(VGPR) or PR per International Myeloma Working Group criteria.sCR: CR& normal serum free light chain(sFLC)ratio &absence of clonal cells in BMB/BMA by immunohistochemistry, immunofluorescence or flow cytometry.CR: negative immunofixation on serum &urine, disappearance of soft tissue plasmacytoma &<5% plasma cells in BMA, if disease measured by sFLC only,preceding criteria plus normal sFLC ratio.VGPR:Serum & urine M-protein detectable by immunofixation but not on electrophoresis; or >=90% reduction in serum&urine M-protein level <100mg/24h.PR:>=50% reduction in serum M-protein & reduction in 24h urinary M-protein by >=90% or <200 mg/24h. If serum & urine M-protein unmeasurable,VGPR & PR: >=90% &>=50% decrease in difference respectively between involved & uninvolved sFLC levels & if present at baseline,>=90% & >=50% reduction in soft tissue plasmacytomas' size.
Time Frame: From date of first dose until confirmed disease progression, death, start of new anticancer therapy, whichever occurred first (maximum of 65.1 weeks of treatment)
Population: SAS included all enrolled participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Percentage of participants | 50.0 [6.8 to 93.2]

14. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined for participants with confirmed objective response (sCR,CR,VGPR and PR) as the time from first date of study intervention to the date of first documentation of objective response. sCR: CR and normal sFLC ratio with absence of clonal cells in BMB/BMA by immunohistochemistry, immunofluorescence or flow cytometry.CR: negative immunofixation on serum and urine,disappearance of soft tissue plasmacytoma, <5% plasma cells in BMA, if disease measured by sFLC only,preceding criteria plus normal sFLC ratio.VGPR:Serum and urine M-protein detectable by immunofixation but not on electrophoresis; or >=90% reduction in serum and urine M-protein level <100mg/24h.PR:>=50% reduction in serum M-protein and reduction in 24h urinary M-protein by >=90% or <200 mg/24h.If serum and urine M-protein unmeasurable,VGPR & PR: >=90%,>=50% decrease in difference respectively between involved and uninvolved sFLC levels,if present at baseline,>=90%, >=50% reduction in soft tissue plasmacytomas' size.
Time Frame: From date of first dose to the first documentation of objective response that is subsequently confirmed (maximum of 65.1 weeks of treatment)
Population: SAS included all enrolled participants who received at least 1 dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Elranatamab
Number analyzed (Participants) | 2
Months | 1.396 [1.18 to 1.61]

15. Secondary Outcome: Duration of Response (DOR)
Description: DOR: time from first documentation of objective response subsequently confirmed, until first documentation of confirmed PD or death due to any cause, whichever occurred first. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5g/dL]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200mg/24h]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved sFLC levels [absolute increase >10mg/dL]; in participants without measurable serum, urine M-protein levels & involved sFLC levels: bone marrow plasma-cell % irrespective of baseline status [absolute increase >=10%]; appearance of new lesion,>=50% increase from nadir in SPD of >1 lesion, or >=50% increase in longest diameter of previous lesion >1cm in short axis; >=50% increase in circulating plasma cells [>=200cells/μL] if this is the only measure of disease.
Time Frame: From first documentation of objective response subsequently confirmed until confirmed PD or death due to any cause, or start of new anticancer therapy, whichever occurs first, or censoring date (maximum of 65.1 weeks of treatment)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Elranatamab
Number analyzed (Participants) | 2
Months | 12.70 [10.4 to NA] — Upper limit could not be estimated due to insufficient number of participants with the event.

16. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) was the time from the first date of the study intervention to the date of the first documentation of confirmed progression, or death due to any cause.
Time Frame: From date of first dose until confirmed PD or death due to any cause, or start of new anticancer therapy, whichever occurs first, or censoring date (maximum of 65.1 weeks of treatment)
Population: SAS included all enrolled participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Months | NA [NA to NA] — Data for PFS was not planned to be summarized per Statistical Analysis Plan (SAP). Individual data was collected but not reported as it would lead to re-identification of participants.

17. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was the time from the first date of the study intervention to the date of death due to any cause. Participants not known to have died are censored on the date of last known alive.
Time Frame: From the date of first dose until death due to any cause or censoring date (maximum of 65.1 weeks of treatment)
Population: SAS included all enrolled participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Months | NA [NA to NA] — Data for OS was not planned to be summarized per SAP. Individual data was collected but not reported as it would lead to re-identification of participants.

18. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: MRD negativity rate was defined as percentage of participants with CR or sCR with negative MRD per IMWG sequencing criteria by bone marrow aspirate (BMA). sCR: CR and normal sFLC ratio with absence of clonal cells in BMB/BMA by immunohistochemistry, immunofluorescence or flow cytometry.CR: negative immunofixation on serum and urine, disappearance of soft tissue plasmacytoma and <5% plasma cells in BMA, if disease measured by sFLC only, preceding criteria plus normal sFLC ratio. MRD was reported at threshold frequency of 10^5 and 10^6.
Time Frame: as for outcome 13
Population: SAS included all enrolled participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Elranatamab
Number analyzed (Participants) | 4
Percentage of participants
  Threshold: 10^5 | 25.0 [0.63 to 80.59]
  Threshold: 10^6 | 25.0 [0.63 to 80.59]

ADVERSE EVENTS:
Time Frame: From first dose of study intervention and up to 90 days after last dose or start of new anticancer therapy (maximum of 65.1 weeks of treatment)
Description: Same event may appear as both SAE and non-SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety analysis set evaluated. All-Cause Mortality: the total number of deaths during study, from first dose and up to the end of the study are reported for all treated participants and includes deaths which occurred after 90 days post last dose of study intervention.
Arm/Group | Elranatamab
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elranatamab (N=4)
Death (General disorders) | 1
Malaise (General disorders) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elranatamab (N=4)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 3
Vertigo (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Injection site reaction (General disorders) | 2
Pyrexia (General disorders) | 2
Cytokine release syndrome (Immune system disorders) | 4
Hypogammaglobulinaemia (Immune system disorders) | 2
Bronchitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Insomnia (Psychiatric disorders) | 1
Pneumonia (Infections and infestations) | 3
Tooth loss (Gastrointestinal disorders) | 1
Weight decreased (Investigations) | 2
Wound (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to character limitation in outcome measure(OM)description, expanded form for ICANS, ASTCT, ICE is provided here. Immune Effector Cell-Associated Neurotoxicity, American Society for Transplantation and Cellular Therapy, Immune Effector Cell-Associated Encephalopathy respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT04798586/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT04798586/SAP_001.pdf